CLINICAL TRIAL: NCT04088006
Title: A Prospective, Monocentric, Intra-individual, Randomized Clinical Investigation to Evaluate the Efficacy and Safety of Stylage® HydroMax on Skin Moisturization and Elasticity
Brief Title: The Evaluation of Efficacy and Safety of Hyaluronic Acid Injection on Skin Moisturization and Elasticity
Acronym: HYDRELA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-A02934-51
Record Dates: First submitted 2019-09-06; First posted 2019-09-12 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Aging
Keywords: Aging; Skin dryness; Skin elasticity; Hyaluronic acid; Injection; Cheek; Neckline area; Healthy subjects; Intra-individual; Independent evaluators; Prospective; Randomized study

STUDY DESIGN:
Intervention Model Description: Intra-individual study with treatment of one cheek and one side of neckline area per subject in a randomly fashion.
  Variation of moisturization, elasticity and roughness between treated areas and non-treated areas of each subject measured at different study timepoints.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Subjects and injectors will be unblinded. All investigators in charge of clinical examination and assessment of local tolerance, as well as all technicians in charge of measurements of moisturization, elasticity, roughness and management of subject questionnaire will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated cheek and neckline area (Experimental): Intra-individual study with one cheek and one side of neckline area treated
  Interventions: Device: Injection of STYLAGE® HydroMax
- Non-treated cheek and neckline area (No Intervention): Intra-individual study with one cheek and one side of neckline area non-treated

INTERVENTIONS:
Device: Injection of STYLAGE® HydroMax — STYLAGE® HydroMax is a hyaluronic acid injectable gel intended to improve skin moisturization and elasticity of the face and neckline area in this study.
  A total of 3 injection sessions will be performed one month apart for each subject.
  At each injection session, 1 mL of product will be injected in the mid to deep dermis of one cheek and another 1 mL in one site of neckline area for each subject.
  Other Names: Injection of hyaluronic acid gel
  Arms: Treated cheek and neckline area

SUMMARY:
STYLAGE® HydroMax is a CE-marketed hyaluronic acid gel intended to improve skin moisturization and elasticity through injection into the dermis of the face, neck, neckline area and back of the hand. In this study, 47 female healthy subjects between the ages of 35 and 65, who have signs of cutaneous dryness and lack of elasticity on the cheek and on the neckline area, who have given her informed consent and met all the eligibility criteria, will be enrolled. One month apart subjects will randomly receive 3 injections of product in one cheek and in one side of the neckline area. Subjects will come to a total of 8 visits over a period of 9 months. Variation of moisturization, elasticity and roughness of treated areas in comparison with non-treated areas will be measured using specific devices by independent evaluators. Global aesthetic improvement, subject satisfaction, pain at injection and safety will also be assessed.

DETAILED DESCRIPTION:
This is a prospective, single center, randomized, intra-individual study with blinded evaluators assessing the efficacy and safety of STYLAGE® HydroMax on skin moisturization and elasticity on the cheek and neckline area. Forty seven female subjects will be enrolled and will receive 3 injections of product one month apart on the cheek and neckline area in a randomized fashion with the contralateral non-treated cheek and neckline area. Injection will be performed into the mid to deep dermis of the cheek and neckline area (1 mL per session and per area) by micro-papular injection technique. Subjects will be followed up at 1, 2, 3, 4, 6 and 9 months timepoints. Variation of moisturization, elasticity and roughness of treated areas in comparison with non-treated areas will be measured using Corneometer®, Cutometer®, Dermatop® or Primos Lite® respectively. Global aesthetic improvement, subject satisfaction, pain at injection and safety will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject.
* Female between 35 and 65 years.
* Having given freely and expressly her informed consent.
* With signs of cutaneous dryness on the cheeks and neckline area (checked by measurements using Corneometer® <60 arbitrary unit (AU) on each cheek).
* With signs of a mild to moderate lack of elasticity on face and neckline area following investigator assessment.
* Psychologically able to understand the study related information and to give a written informed consent.
* Affiliated to a health social security system.
* Female of childbearing potential should use a medically accepted contraceptive regimen since at least 12 weeks before the beginning of the study and during all the study.
* Agreeing not to change any hormonal treatment (including contraceptive treatment) during the whole study.
* Agreeing to keep their usual cleansing / care products during the whole study period.
* Agreeing to apply a sun protection factor SFP50 cream during non-intensive exposure to sunlight.

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the study.
* With a tattoo, a scar, moles, too many hairs or anything on the studied zones which might interfere with the evaluation.
* Who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* In a social or sanitary establishment.
* Having received 4500 euros indemnities for participation in researches involving human beings in the 12 previous months, including participation in the present study.
* Participating to another research on human beings or who is in an exclusion period of one.
* Intensive exposure to sunlight or UV-rays within the previous month and foreseen during the study.
* Suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results.
* With known history of or suffering from autoimmune disease and/or immune deficiency.
* Suffering from inflammatory and/or infectious cutaneous disorders in or near the studied zones (herpes, acne, mycosis, papilloma…). Subject with recurrent herpes is not eligible even if asymptomatic at time of inclusion.
* Having history of severe allergy or anaphylactic shock including hypersensitivity to hyaluronic acid or to one of the component of the tested device, antiseptic solution or anaesthesia product if applicable.
* With fructose intolerance.
* With a past history of streptococcal disease, such as acute rheumatic fever or recurrent sore throats.
* Predisposed to keloids or hypertrophic scarring.
* Prone to develop inflammatory skin conditions or having tendency to bleeding disorders.
* Having received treatment with a laser, a dermabrasion, a surgery, a deep chemical peeling or other ablative procedure on the cheeks or the neckline area within the past 12 months prior to study start.
* Having received injection with a resorbable filling product in the cheeks or the neckline area within the past 18 months prior to study start.
* Having received at any time injection with a slowly resorbable filling product (polylactic acid, calcium hydroxyapatite, combinations of hyaluronic acid (HA) and hypromellose, HA and dextran microbeads or HA and TriCalcium Phosphate (TCP), …) or with a non-resorbable filling product (polyacrylamide, silicone, combination of methacrylic polymers and collagen, polymer particles, …).
* Having received at any time a treatment with tensor threads on the face or the neckline area.
* Having started or changed her oral contraceptive or any other hormonal treatment during 12 weeks prior to study start.
* Using medication such as aspirin, NSAIDs (ibuprofen, naproxen, …), antiplatelet agents, anticoagulants, vitamin C within one week prior to study start and agreeing not to take such treatments within 1 week prior to the second and third injections or being a chronic user.
* Undergoing a topical treatment on the test area or a systemic treatment:

  * anti-histamines during the 2 weeks prior to study start;
  * immunosuppressors and/or corticoids during the 4 weeks prior to study start;
  * retinoids during the 6 months prior to study start.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Variation of cheek cutaneous moisturization | Month 3
  Variation from baseline before treatment (D0) to 3 months after treatment initiation of the cutaneous moisturization on the cheek, in comparison with the non-treated cheek, by an independent evaluator using Corneometer®.

SECONDARY OUTCOMES:
Variation of cheek cutaneous moisturization | Month 1, Month 2, Month 4, Month 6, Month 9
  Variation from baseline to 1, 2, 4, 6 and 9 months after treatment initiation of the cutaneous moisturization on the cheek in comparison with the non-treated cheek by a blinded independent evaluator using Corneometer®.
Variation of neckline area cutaneous moisturization | Month 1, Month 2, Month 3, Month 4, Month 6, Month 9
  Variation from baseline to 1, 2, 3, 4, 6 and 9 months after treatment initiation of the cutaneous moisturization on the neckline area in comparison with the non-treated neckline area by a blinded independent evaluator using Corneometer®.
Variation of cheek and neckline area cutaneous elasticity | Month 1, Month 2, Month 3, Month 4, Month 6, Month 9
  Variation from baseline to 1, 2, 3, 4, 6 and 9 months after treatment initiation of the cutaneous elasticity on the cheek and neckline area in comparison with the non-treated cheek and neckline area by a blinded independent evaluator using Cutometer®.
Variation of cheek cutaneous roughness | Month 1, Month 2, Month 3, Month 4, Month 6, Month 9
  Variation from baseline to 1, 2, 3, 4, 6 and 9 months after treatment initiation of the cutaneous roughness on the cheek in comparison with the non-treated cheek by a blinded independent evaluator using Dermatop®.
Variation of neckline area cutaneous roughness | Month 1, Month 2, Month 3, Month 4, Month 6, Month 9
  Variation from baseline to 1, 2, 3, 4, 6 and 9 months after treatment initiation of the cutaneous roughness on the neckline area in comparison with the non-treated neckline area by a blinded independent evaluator using Primos Lite®.
Evaluation of global aesthetic improvement | Month 1, Month 2, Month 3, Month 4, Month 6, Month 9
  Evaluation by the subject and by the blinded independent evaluator of the global aesthetic improvement of treated and non-treated zones 1, 2, 3, 4, 6 and 9 months after treatment initiation using the Global Aesthetic Improvement Scale (GAIS). The Global Aesthetic Improvement Scale is a 5-score scale (from score 1 to score 5) with minimum scores representing a better outcome. Score 1 corresponds to "Very much improved", score 2 to "Much improved", score 3 to "Improved", score 4 to "No change" and score 5 to "Worse".
Evaluation of subject's satisfaction | Month 1, Month 2, Month 3, Month 4, Month 6, Month 9
  Evaluation of subject's satisfaction 1, 2, 3, 4, 6 and 9 months after treatment initiation using a questionnaire.
Evaluation of pain during injection | Day 0, Month 1, Month 2
  Evaluation of the pain during injection by the subject using a numerical rating scale from 0 to 10.
Report of adverse events | Up to Month 9
  Evaluation of product tolerance by collection of adverse events assessed by subject and independent evaluator.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie CONVERSET-VIETHEL, MD, Principal Investigator
Locations (1):
- Laboratoire DERMSCAN, Villeurbanne, Rhône, France

IPD SHARING:
Plan to Share IPD: No